CLINICAL TRIAL: NCT07228455
Title: The Effect of Humeral Head Depressor Strengthening in Individuals With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Utku Kurtaran, Principal Investigator, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/115-1751
Record Dates: First submitted 2025-09-29; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Participants were quasi-randomly and sequentially assigned to either an intervention group receiving humeral head depressor exercises or a control group receiving routine exercise therapy. Each group followed their respective program for the duration of the study.
Who Masked: Participant
Masking Description: Participants were blinded to their group assignment, but therapist were aware of the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention Group (Experimental): The Intervention group underwent a progressive resistance exercise program to strengthen the humeral head depressors and peri-articular muscles, including the rotator cuff. The exercises were performed 3 times per week for 6 weeks, with each session lasting approximately 1 hour
  Interventions: Behavioral: Humeral Head Depressor Exercises
- The Control Group (Active Comparator): Participants in the control group received standard physical therapy and rehabilitation as usually applied in routine care. Sessions were performed 3 times per week for 6 weeks, each lasting approximately 1 hour.
  Interventions: Behavioral: Standard physical therapy

INTERVENTIONS:
Behavioral: Humeral Head Depressor Exercises — The Intervention group underwent a progressive resistance exercise program to strengthen the humeral head depressors and peri-articular muscles, including the rotator cuff. Exercises were performed 3 times per week for 6 weeks, each session lasting approximately 1 hour
  Arms: The Intervention Group
Behavioral: Standard physical therapy — Participants in this group received standard physical therapy and rehabilitation as usually applied in routine care. Exercises were performed 3 times per week for 6 weeks, each session lasting approximately 1 hour. Outcomes were measured at the same time points as the intervention group.
  Arms: The Control Group

SUMMARY:
Subacromial impingement syndrome is a common musculoskeletal disorder. Therefore, to improve the shoulder biomechanics affected by the syndrome, an intervention group was compared with a control group. The exercise program applied to the intervention group is expected to improve the function of the shoulder complex.

DETAILED DESCRIPTION:
Subacromial Impingement Syndrome (SIS) is one of the most common musculoskeletal problems in the shoulder joint. This study aimed to investigate the effectiveness of a rehabilitation program targeting humeral head depressor muscles on symptoms in individuals with SIS.Participants were randomly divided into study and control groups.Volunteers who complained of shoulder pain for more than a month, who had limitation in passive movement compared to the other side shoulder, who had Neer impingement test, Hawkins test, Jobe supraspinatus test, and who were able to com-municate were included in the study. Individuals 1) Having any neurological condition affecting the upper extremity, 2) having neurological findings related to cervical disc herniation, 3) having a full-thickness rupture of one of the rotator cuff tendons, 4) having calcific tendonitis, 5) having undergone previous shoulder surgery and 6) Physical therapy-rehabilitation for the shoulder with the same complaints in the last 6 months, or 7) receiving corticosteroid injection were excluded from the study. While the control group received standard physical therapy and rehabilitation, the study group underwent a progressive resistance exercise program to strengthen the humeral head depressors and peri-articular muscles, including the rotator cuff. Acromio-humeral distance (AHD) and tendon thickness measurements were evaluated by ultrasonography, while pain intensity was measured through VAS and McGill Questionnaire, upper extremity disability through DASH-T, and kinesiophobia through Fear Avoidance Beliefs Questionnaire, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who complained of shoulder pain for more than a month,
* Who had limitation in passive movement compared to the other side shoulder,
* Who had Neer impingement test, Hawkins test, Jobe supraspinatus test, and -
* Who were able to com-municate were included in the study

Exclusion Criteria:

* Having any neurological condition affecting the upper extremity,
* Having neuro-logical findings related to cervical disc herniation,
* Having a full-thickness rupture of one of the rotator cuff tendons,
* Having calcific tendonitis,
* Having undergone previous shoulder surgery,
* Physical therapy-rehabilitation for the shoulder with the same complaints in the last 6 months,
* Receiving corticosteroid injection were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Acromio-humeral Distance (Ultrasonography, USG) | Baseline and 6 weeks

SECONDARY OUTCOMES:
Tendon Thickness Measurment | Baseline and 6 week
  Supraspinatus Tendon, Infraspinatus Tendon, subscapularis Tendon, Teres Minor Tendon, Long Head Biceps Tendon, Rotator Cuff group Tendons General Thicknesses were evaluated in all planes, by USG using a GE LogiqP6 Pro device and a linear transducer. Imaging was performed using standard shoulder sections while the patients were in a sitting position
Pain (Visual Analog Scale, VAS) | Baseline and 6 weeks
  Pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Pain (McGill Pain Questionnaire-Pain Rating Index) | Baseline and 6 weeks
  Pain will be assessed using the McGill Pain Questionnaire, specifically the Pain Rating Index (PRI). The total score ranges from 0 to 78, with higher scores indicating more severe pain.
Kinesiophobia (Fear Avoidance Beliefs Questionnaire - FABQ, Physical Activity subscale) | Baseline and 6 weeks
  Kinesiophobia will be assessed using the Fear Avoidance Beliefs Questionnaire (FABQ) - Physical Activity subscale (items 2-5). Score range: 0 to 24 (higher scores indicate greater fear-avoidance beliefs related to physical activity).
  Time Frame: Baseline and 6 weeks.
Kinesiophobia (Fear Avoidance Beliefs Questionnaire - FABQ, Work subscale) | Baseline and 6 weeks.
  Kinesiophobia will also be assessed using the FABQ - Work subscale (items 6, 7, 9-12, 15). Score range: 0 to 42 (higher scores indicate greater fear-avoidance beliefs related to work).
Upper Extremity Disability Through (DASH-T) | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet OZGUL, Prof., Principal Investigator — Department of Physical Medicine and Rehabilitation, Kyrenia University Hospital, Kyrenia, Cyprus
Locations (1):
- Near East University Hospital, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
The individual participant data from this study will not be shared.

REFERENCES:
- [Derived] Kurtaran U, Yerlikaya T, Yenen B, Ozgul A. The Effect of Humeral Head Depressor Strengthening on Individuals with Subacromial Impingement Syndrome. Medicina (Kaunas). 2025 Nov 19;61(11):2061. doi: 10.3390/medicina61112061. PMID 41303896